CLINICAL TRIAL: NCT04272411
Title: Effects of Burst and Tonic Spinal Cord Stimulation (SCS) in Chronic Neuropathic Pain on Blood Glucose Levels
Brief Title: SCS Stimulation Clamp to Assess Impact of Stimulation on Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 202/2019BO2
Record Dates: First submitted 2020-02-07; First posted 2020-02-17 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Spinal Cord Stimulation (SCS); Blood Glucose Metabolism; Euglycemic Hyperinsulinemic Clamp

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham SCS stimulation (Sham Comparator): Sham SCS stimulation via implanted neuromodulation device
  Interventions: Device: Sham SCS stimulation
- Tonic SCS stimulation (Active Comparator): Tonic SCS stimulation via implanted neuromodulation device
  Interventions: Device: Tonic SCS stimulation
- Burst SCS Stimulation (Active Comparator): Burst SCS stimulation via implanted neuromodulation device
  Interventions: Device: Burst SCS Stimulation

INTERVENTIONS:
Device: Sham SCS stimulation — Sham SCS stimulation via implanted neuromodulation device for 45 min during the steady state of a hyperinsulinemic euglycemic clamp.
  Arms: Sham SCS stimulation
Device: Tonic SCS stimulation — Tonic SCS stimulation via implanted neuromodulation device for 45 min during the steady state of a hyperinsulinemic euglycemic clamp.
  Arms: Tonic SCS stimulation
Device: Burst SCS Stimulation — Burst SCS stimulation via implanted neuromodulation device for 45 min during the steady state of a hyperinsulinemic euglycemic clamp.
  Arms: Burst SCS Stimulation

SUMMARY:
In 1967 spinal cord stimulation (SCS) for the treatment of chronic neuropathic pain was established. Today various pain syndromes like the failed back surgery syndrome (FBSS), the complex regional pain syndrome (CRPS), ischemic pain or phantom limb pain are treated with SCS. The development of this technique based on the so called "Gate Control Theory" which states that stimulation of the mechanosensitive Aβ fibers suppresses the transmission of pain stimuli via the pain-sensitive C fibers to the brain in the spinal cord. Conventional SCS consists of periodically emitted tonic stimuli with a frequency between 30 and 120 Hz. During implantation, the electrodes are placed in the epidural space in such a way that the paraesthesia caused by nerve stimulation covers the painful area (dermatome), thus relieving the pain. In 2010 de Ridder et al. published an article presenting the so called "Burst Stimulation" where series of high-frequency impulses are released at defined time intervals (frequency: 40 Hz with peaks of 500 Hz per volley). Compared to the tonic SCS the burst technique is more effective and in most cases no paraesthesia is reported. However, potential effects of SCS stimulation on other organ systems have only been insufficiently examined.Especially possible effects of SCS on the glucose metabolism has not been investigated so far. However, it is important to investigate a possible effect for two reasons: SCS could cause severe hypoglycemia which must be avoided. Furthermore, if SCS affects blood sugar levels, it is also of interest what mechanisms are involved and how this knowledge can be used to control elevated blood glucose levels.

The present study is a pilot. The investigators want to examine possible effects of SCS therapy on blood glucose metabolism. Therefore hyperinsulinemic euglycemic clamps with an insulin infusion of 1mU / kg body weight per minute are performed. During the clamp the investigators apply different SCS techniques in a randomly order. Insulinsensitivity is determined at different time points.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures.
* HbA1c < 6,0%
* state after implantation of an neuromodulation device
* Clinical routine blood parameters within the normal ranges

Exclusion Criteria:

* diabetes mellitus
* Acute diseases such as infections (e.g.) within the last four weeks
* Hb < 13 g/dl
* anamnestic heparin-induced thrombocytopenia
* any neurologic or psychiatric disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in peripheral insulin sensitivity (tonic/burst versus sham stimulation) | 130-150 minutes, 190-210 minutes and 250-270 minutes respectively during euglycemic clamp
  Effect of tonic or burst versus sham SCS stimulation on insulin sensitivity assessed by hyperinsulinemic euglycemic clamp.

SECONDARY OUTCOMES:
Change in peripheral insulin sensitivity (tonic versus burst stimulation) | 130-150 minutes, 190-210 minutes and 250-270 minutes respectively during euglycemic clamp
  Differential effects of tonic versus burst SCS stimulation on insulin sensitivity assessed by hyperinsulinemic euglycemic clamp.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hopsital Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No